CLINICAL TRIAL: NCT04452162
Title: Physiologic MR Imaging in Distinguishing Benign From Malignant Salivary Gland Tumors
Brief Title: Physiologic MR Imaging of Salivary Gland Tumors
Acronym: PSGT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: McCabe Fund (Unknown)
Responsible Party: Principal Investigator, Sanjeev Chawla, Assistant Research Professor of Radiology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25319; 834242 (Other: IRB)
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Salivary Gland Tumor
MeSH Terms: conditions — Salivary Gland Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Salivary Gland Tumor (Other)
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — You are being asked to complete one research MRI scan with and without contrast since your most recent clinical evaluation and/or prior imaging has shown the presence of a suspicious salivary gland tumor, prior to your scheduled upcoming surgery. MRI contrast agents act like a dye to make MRI pictures brighter and easier to read. During each MRI scan, you will have an intravenous line (IV line) placed. The IV line allows the contrast agent to be injected into your vein. If you have a history of renal disease you may be asked to complete a blood draw of approximately 2.5cc (½ teaspoon), for glomerular filtration rate (GFR) assessment for participation into the study.

SUMMARY:
The goal of this study is to use advanced Magnetic Resonance Imaging (MRI) techniques to help identify the difference between cancerous and non-cancerous salivary gland tumors for improving treatment strategies and to aid in the prediction of disease progression.

DETAILED DESCRIPTION:
The goal of this proposed study is to investigate the potential utility of combined analysis of parameters (Ktrans, ti and ADC) in discriminating benign from malignant salivary glands tumors (SGTs). A total of 30 treatment naïve patients suspicious of SGT as observed on clinical evaluation and prior routine CT, MRI, Ultrasound, FNAC and/or PET will undergo 3T MRI. The MRI protocol will include acquisition of anatomical images with and without contrast agent injection, diffusion imaging and dynamic contrast enhanced-MRI.

ELIGIBILITY:
Inclusion Criteria:

* Possess a salivary gland lesion of 1cm3 size
* Have no prior history of treatment for salivary gland lesion

Exclusion Criteria:

* Has any prior history of cancer other than SGT
* Has any MRI contra-indications
* Has a history of known renal disease.
* Has history of prior radiation to head and neck region
* Is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Differentiation and Progression Free | 6 Month after the end of treatment
  Differentiation of malignant from benign neoplasms and progression free survival at 6 month starting from end of chemo-radiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Chawla, Principal Investigator — Professor
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No